CLINICAL TRIAL: NCT01133535
Title: The IRAP Registry is a Multi-center Prospective, Collaborative Database Designed to Create a National Registry That Collects Information Concerning Episodes of Idiopathic Recurrent Acute Pancreatitis From Major 'Pancreas' Centers. Intent is to do a Comparative Effectiveness Study of Interventions.
Brief Title: Idiopathic Recurrent Acute Pancreatitis (IRAP)
Acronym: IRAP
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: AHC-001
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2014-06

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pancreatitis, acute, recurrent: Patients with acute recurrent pancreatitis where the cause is unknown

SUMMARY:
The purpose of this study is to collect standardized data on the diagnosis and management of idiopathic (unknown cause) recurrent acute pancreatitis. The intent is to collect data for at least five years to obtain information regarding long-term outcomes and obtain comparative effectiveness data.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Able to provide consent
3. More than one documented episode of pancreatitis (>3 fold elevation of amylase and or lipase with abdominal pain or with body imaging consistent with pancreatitis: need two of the three)
4. Subjects with abdominal pain and enzyme elevation which is <3 fold above normal or absence of imaging findings: these subjects who are undergoing endoscopic interventions but do not fit the "classic criteria" for pancreatitis will be included but the analysis of data of these subjects would be done separately.

Note: subjects with a diagnosis of pancreas divisum and or Sphincter of Oddi dysfunction diagnosed prior to or after entry into the study will be included in the study but their data will be analyzed separately because of the controversy regarding the association of these entities with pancreatitis.

Exclusion Criteria:

1. Unable to give informed consent.
2. Definite evidence of biliary or alcoholic pancreatitis.
3. Clear evidence of hypertriglyceridemia-induced pancreatitis (triglycerides >1,000 mg/dl).
4. Post-ERCP pancreatitis, drug-induced pancreatitis, or any identifiable cause for pancreatitis.
5. History of pancreatic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with recurrent pancreatitis presenting to major centers for pancreatic disorders
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
IDIOPATHIC RECURRENT ACUTE PANCREATITIS (IRAP) | The goal is to recruit 1000 subjects in 5 years.
  Expect 750 to be treated with ERCP Expect 250 to be treated with conservative treatment. Therefore, the smaller group was used for the sample size analysis.
  Smallest difference in QOL for treatment is expected to be 10-20%. For smaller of two treatment groups (N=250), no effect would be 0 got better and 250 did not. If 10% of the subjects improved, 25 would get better and 225 would not. Result: Chi-square analysis yielded a highly significantly difference as follows. Chi-square= 24.253 with 1 degrees of freedom. (P = <0.001). Yates correction for continuity was used in calculating this test.An alternate analysis is that for no effect, 125 subjects would get better and 125 patients would not (random effects model).

CONTACTS AND LOCATIONS:
Overall Officials: Nalini M Guda, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora St. Lukes Medical Center of Aurora Health Care, Milwaukee, Wisconsin, United States